CLINICAL TRIAL: NCT04547309
Title: Research for the Molecular Imaging of the HER2 Targeting Tracer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); North Sichuan Medical College (Other)
Responsible Party: Principal Investigator, Hua Zhu, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018KT61/2019KT114
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-08

CONDITIONS: HER2 Positive or Suspicious Positive Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga/18F-HER2 Affibody PET/CT scan (Experimental)
  Interventions: Radiation: 68Ga/18F-HER2 Affibody PET/CT scan

INTERVENTIONS:
Radiation: 68Ga/18F-HER2 Affibody PET/CT scan — HER2 Affibody, labeled with PET radio-nuclide ( 68Ga or F-18) will be used as a molecular imaging tracer for PET/CT scan. All participants will undergo 68Ga/18F-HER2 Affibody PET/CT scan.

SUMMARY:
To use the molecular PET radionuclide (Ga-68 or F-18) labelled HER2 Affibody to detect the expression of HER2 in the primary and metastatic lesions in patients with HER2 positive or suspicious positive tumors; to detect the expression heterogeneity of HER2 in the lesions and inter-lesions; to observe the change of HER2 expression in the course of treatment. To provide an approach for screening patients high expression of HER2, efficacy monitoring, drug resistance and early warning of recurrence and metastasis to achieve the individualized antitumor treatment of targeted drugs.

DETAILED DESCRIPTION:
HER2 is an important biomarker and directly inﬂuences the treatment effect. The guidelines indicate that only HER2-positive patients are eligible for trastuzumab therapy.HER2 positivity is defined as a HER2 score of 3+ by IHC or FISH. However, gastroscopic biopsies are spatiotemporally limited because of the highly heterogeneous expression of HER2. And this procedure is invasive and may substantially increase the incidence of side effects. Additionally, patients with false-negative HER2 results miss the chance for targeted therapy. Moreover, HER2 status can change during the disease process.Thus, a noninvasive, whole-body, HER2-targeted imaging method may be valuable for choosing patients suitable for anti-HER2 therapy and monitoring the therapeutic efficacy. Direct labeling of HER2 antibodies with radionuclides allows clinicians to monitor HER2-targeted therapy and assists in patient staging. With the feasibility of a long half-life and decay time, positron emission tomography (PET) nuclides, such as 64Cu (T1/2= 12.7 h) and 89Zr (T1/2= 78.4 h), can label trastuzumab for the clinical PET imaging of HER2 in GC and breast cancer. Because of the long half-life of 89Zr, 89Zr-trastuzumab is estimated to produce a dosimetry exposure of 0.5 mSv/MBq (compared with the 0.019 mSv/MBq of 18FDG) in patients. Additionally, imaging needs to be performed several days after injection due to the slow blood clearance of antibodies.

In this study, 68Ga-HER2 Affibody or 18F-HER2 Affibody PET/CT imaging will be performed in patients with HER2-positive tumors to access the potential of 68Ga-HER2 Affibody or 18F-HER2 Affibody PET/CT to screen patients who can benefit from HER2 target treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged > 18 years old; ECOG 0 or 1;
2. Patients with HER2 positive or suspicious positive tumors;
3. Has at least one measurable target lesion according to CT or MRI;
4. Life expectancy ≥ 12 weeks.

Exclusion Criteria:

1. Significant hepatic or renal dysfunction;
2. Is pregnant or ready to pregnant;
3. Cannot keep their states for half an hour;
4. Refused to join the clinical research;
5. Suffering from claustrophobia or other mental disorders;
6. Any other situation that researchers considered it unsuitable to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
SUV | 3 years
  The uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value (SUV) on PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Hua Zhu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo X, Liu J, Ma H, Ma X, Liang X, Zhu H, Li C, Yang Z, Zhou N. Al 18 F-NOTA-HER2-BCH Versus 18 F-FDG PET/CT for Detecting Bone Metastases : Sensitivity and Quantitative Comparison. Clin Nucl Med. 2026 Feb 1;51(2):123-131. doi: 10.1097/RLU.0000000000006249. Epub 2025 Dec 22. PMID 41474774
- [Derived] Guo X, Liu J, Lin S, Gui X, Ding J, Liu T, Zhou N, Li S, Zhu H, Yang Z. Detectability of Al 18 F-NOTA-HER2-BCH PET for Nodal Metastases in Patients With HER2-Positive Breast Cancer. Clin Nucl Med. 2025 May 1;50(5):381-387. doi: 10.1097/RLU.0000000000005686. Epub 2025 Jan 24. PMID 39854676
- [Derived] Gui X, Liang X, Guo X, Yang Z, Song G. Impact of HER2-targeted PET/CT imaging in patients with breast cancer and therapeutic response monitoring. Oncologist. 2025 Jan 17;30(1):oyae188. doi: 10.1093/oncolo/oyae188. PMID 39083323
- [Derived] Guo X, Zhou N, Liu J, Ding J, Liu T, Song G, Zhu H, Yang Z. Comparison of an Affibody-based Molecular Probe and 18F-FDG for Detecting HER2-Positive Breast Cancer at PET/CT. Radiology. 2024 Jun;311(3):e232209. doi: 10.1148/radiol.232209. PMID 38888484